CLINICAL TRIAL: NCT01662817
Title: Effectiveness of Physicians' Education, Implementation and Follow up of Current Recommendations Regarding Screening for Major Depressive Disorder in High Risk Patients on Improving the Under-Recognition Rates of Depression in Primary Care
Brief Title: Major Depressive Disorder (MDD)
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 13487; H6U-XM-S007 (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-27; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention: Intervention group primary care physician (PCP) receives one day training in depression screening guidelines and uses guidelines for six months
  Interventions: Behavioral: Intervention
- Control: Control group PCP manages depression in the usual way for six months
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — PCP receives one day training in depression screening guidelines and uses guidelines for six months
  Groups: Intervention
Behavioral: Control — PCP manages depression in the usual way for six months
  Groups: Control

SUMMARY:
The purpose of this study is to assess the effectiveness of systematic screening for depression in high-risk patient participants in everyday clinical practice. Systematic screening for depression in high-risk patients is recommended to be included as a usual practice but its effectiveness in this context remains controversial. In this study, 35 primary care physicians (PCPs) in Spain were assigned to intervention (receive one day training in depression screening guidelines and use guidelines for six months) and 34 PCPs were assigned to a control group (manage depression in the usual way for six months). There were a total of 525 patient participants with MDD.

ELIGIBILITY:
Inclusion Criteria:

* PCP Participants: PCPs informed of the study design and who agreed to be randomized to the intervention or control group
* Patient Participants: Aged 18 years or older who provide a written consent for the collection and use of their clinical data

Exclusion Criteria:

* PCP Participants: If they already follow the recommendations on screening or were planning to do so. If they will be absent from their practice for a significant period during the study, or if they do not usually manage depression
* PCP Participants: Those who were not able to understand the aims of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Physicians are given the intervention of education to utilize on screened and consented patient participants under the PCP care.
Sampling Method: Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Patient Participants with Under-Recognized Major Depressive Disorder (MDD) Episodes at 24 Weeks | 24 Weeks

SECONDARY OUTCOMES:
Percentage of Patient Participants with Under-Treatment of MDD Episodes at 24 Weeks | 24 Weeks
Change from Baseline in Primary Care Physician (PCP) Adherence to Intervention Questionnaire at 24 Weeks | Baseline, 24 Weeks
Change from Baseline in PCP Feasibility of Intervention Questionnaire at 24 Weeks | Baseline, 24 Weeks
Change from Baseline in PCP Acceptance of Intervention Questionnaire at 24 Weeks | Baseline, 24 Weeks
Mean Duration of Depressive Episodes in Patient Participants | 24 Weeks
Clinical Global Impressions: Severity (CGI-S) Score in Patient Participants | 24 Weeks
Sheehan Disability Scale (SDS) Score in Patient Participants | 24 Weeks
Mean Duration of Sick Leave Due to Depression in Patient Participants | 24 Weeks
Percentage of Patient Participants with Sick Leave Due to Depression | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid, Spain

REFERENCES:
- [Derived] Romera I, Montejo AL, Aragones E, Arbesu JA, Iglesias-Garcia C, Lopez S, Lozano JA, Pamulapati S, Yruretagoyena B, Gilaberte I. Systematic depression screening in high-risk patients attending primary care: a pragmatic cluster-randomized trial. BMC Psychiatry. 2013 Mar 13;13:83. doi: 10.1186/1471-244X-13-83. PMID 23497463